CLINICAL TRIAL: NCT06473948
Title: A Phase 1, Single Center, Randomized, Double-Blind, Placebo-Controlled, Single-Dose Study to Evaluate the Effect of JMKX001899 on the QTc Interval in Healthy Subjects
Brief Title: To Assess the Effects of Single Dose of JMKX001899 on QTc Interval in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jemincare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: JY-JM1899-106
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Participants will receive JMKX001899 500 once on Day 1
  Interventions: Drug: JMKX001899; Drug: Placebo
- Cohort 2 (Experimental): Participants will receive JMKX001899 750 once on Day 1
  Interventions: Drug: JMKX001899; Drug: Placebo
- Cohort 3 (Experimental): Participants will receive JMKX001899 1000 once on Day 1
  Interventions: Drug: JMKX001899; Drug: Placebo

INTERVENTIONS:
Drug: JMKX001899 — Participants will receive JMKX001899 500mg tablet, orally once on Day 1
  Arms: Cohort 1
Drug: JMKX001899 — Participants will receive JMKX001899 750mg tablet, orally once on Day 1
  Arms: Cohort 2
Drug: JMKX001899 — Participants will receive JMKX001899 1000mg tablet, orally once on Day 1
  Arms: Cohort 3
Drug: Placebo — Participants will receive JMKX001899 matching placebo, tablet, orally once on Day 1

SUMMARY:
Study to assess the effect of JMKX001899 on QTc interval in healthy volunteers

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Placebo-Controlled, Single-Dose Escalation Study to Evaluate the Pharmacokinetics and the Effect on Cardiac Repolarization of JMKX001899 Administered as a Tablet Formulation Under Fed Conditions in Healthy Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, male or female 18-45 years of age, inclusive.
2. Body mass index (BMI) between 19 and 28 kg/m2 (inclusive) and weight at least 50 kg.
3. Participant must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study.

Exclusion Criteria:

1. Patients with a history of clinically significant diseases including, but not limited to, gastrointestinal, renal, liver, neurological, hematological, endocrine, neoplastic, pulmonary, immune, psychiatric, or cardiovascular and cerebrovascular diseases, epilepsy, bipolar disorder/mania, intraocular hypertension, or acute angle-closure glaucoma.
2. Female subjects with a positive pregnancy test or lactating.
3. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) or Treponema pallidum（TP-Ab）

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-07-10 (Estimated); Primary Completion 2024-09-24 (Estimated); Study Completion 2025-02-27 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of a single dose of JMKX001899 on the change in time-matched QTc intervals compared with placebo | 48 hours
  QTc interval was measured by electrocardiograms to evaluate the potential effect of JMKX001899 plasma concentrations on the QTc interval using linear mixed-effect exposure-response modeling, including the predicted ddQTc at Cmax values corresponding to exposure levels

IPD SHARING:
Plan to Share IPD: No